CLINICAL TRIAL: NCT01198366
Title: A Phase II, Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Safety and Immunogenicity of AERAS-402 in BCG-vaccinated, HIV-uninfected Infants Without Evidence of Tuberculosis
Brief Title: Study of AERAS-402 in Healthy Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-029-402
Record Dates: First submitted 2010-09-07; First posted 2010-09-10 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Vaccine; Immunogenicity; Prevention of Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Dose Finding Gr 1 placebo x 2 (Placebo Comparator): Subjects received two doses (x2) of placebo (sterile buffer) on study days 0 and 28.
  Interventions: Biological: Placebo
- Dose Finding Gr 2 AERAS-402 (1.5 x 10^10 vp) x2 (Experimental): Subjects received two doses (x2) of AERAS-402 (1.5 x 10^10 vp) on study days 0 and 28.
  Interventions: Biological: AERAS-402 1.5 x 10^10 vp
- Dose Finding Gr 3 AERAS-402 (3.0 x 10^10 vp) x 2 (Experimental): Subjects received two doses (x2) of AERAS-402 (3.0 x 10^10 vp) on study days 0 and 28.
  Interventions: Biological: AERAS-402 3.0 x 10^10 vp
- Dose Finding Gr 4 AERAS-402 (1.0 x 10^11 vp) x 2 (Experimental): Subjects received two doses (x2) of AERAS-402 (1.0 x 10^11 vp) on study days 0 and 28.
  Interventions: Biological: AERAS-402 1.0 x 10^11 vp
- Expanded Safety Phase Gr 5 AERAS-402 (1.0 X 10^11 vp) x 3 (Experimental): Subjects received 3 doses (x3) of AERAS-402 (1.0 X 10^11 vp) on days 0, 28 and 280.
  Interventions: Biological: AERAS-402 1.5 x 10^10 vp
- Expanded Safety Phase Gr 5 Placebo x3 (Placebo Comparator): Subjects received 3 doses (x3) of placebo (sterile buffer) on days 0, 28 and 280.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AERAS-402 1.5 x 10^10 vp
  Arms: Dose Finding Gr 2 AERAS-402 (1.5 x 10^10 vp) x2; Expanded Safety Phase Gr 5 AERAS-402 (1.0 X 10^11 vp) x 3
Biological: AERAS-402 3.0 x 10^10 vp
  Arms: Dose Finding Gr 3 AERAS-402 (3.0 x 10^10 vp) x 2
Biological: AERAS-402 1.0 x 10^11 vp
  Arms: Dose Finding Gr 4 AERAS-402 (1.0 x 10^11 vp) x 2
Biological: Placebo
  Arms: Dose Finding Gr 1 placebo x 2; Expanded Safety Phase Gr 5 Placebo x3

SUMMARY:
AERAS-402 will be given to infants of at least 16 weeks of age who have already been vaccinated with BCG to determine if AERAS-402 will increase protection of infants to tuberculosis.

DETAILED DESCRIPTION:
The only currently available tuberculosis vaccine, bacillus Calmette-Guérin (BCG), is estimated to reduce the risk of tuberculosis (TB) in children by up to 70-80%, but protection is incomplete. Efforts to increase TB protection in children include new vaccines for primary immunizations as well as combinations of vaccines given as primary and boosting vaccinations.

AERAS 402 is a live recombinant serotype 35 replication deficient adenovirus vector expressing a fusion protein of three Mycobacterium tuberculosis (Mtb) antigens (Ag85A, Ag85B and TB10.4). It presents Mtb antigens in the setting of a new, live, replication-deficient adenovirus vaccine that may increase T cell-mediated immunity and thus protection from tuberculosis. AERAS-402 appears safe and immunogenic in adults. Since BCG-vaccinated infants are the population for which AERAS-402 might be indicated, AERAS-402 will be administered to infants of at least 16 weeks of age who have already been vaccinated with BCG. This is the first Phase II study of AERAS-402 in infants.

ELIGIBILITY:
Inclusion Criteria:

1. Parent/legal guardian has completed the written informed consent process
2. Is age greater than or equal to 112 days (16 weeks) and less than or equal 182 days (26 weeks) on Study Day 0
3. Has general good health, confirmed by medical history and physical examination
4. Is up to date on all Expanded Program of Immunization (EPI) immunizations for his/her age with a minimum of 14 days between the last EPI vaccination and administration of study vaccine on Study Day 0
5. Has ability to complete follow-up period of 728 days as required by the protocol
6. Parent/legal guardian is able and willing to stay in contact with the study site for the duration of the study and to provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study
7. Has completed simultaneous enrollment in Aeras Vaccine Development Registry protocol
8. Had BCG vaccination ≥ 3 months prior to randomization documented by medical card

Exclusion Criteria:

1. Acute illness, evidence of any significant active infection or temperature >=37.5°C on the day of randomization
2. Used immunosuppressive medication within 45 days before entry into the study (inhaled and topical corticosteroids are permitted)
3. Received immunoglobulin or blood products within 45 days before entry into the study
4. Ever received any investigational drug therapy or investigational vaccine
5. History or laboratory evidence of individual immunodeficiency virus (HIV-1) infection
6. History of allergic disease or reactions to any component of the study vaccine
7. Previous medical history that may compromise the safety of the participant in the study
8. Evidence of a new acute illness that may compromise the safety of the participant in the study
9. Inability to discontinue daily medications during the study
10. History or evidence of any systemic disease on physical examination or any acute or chronic illness that may interfere with the evaluation of the safety or immunogenicity of the vaccine, e.g., including masses between the leg and abdomen (e.g., inguinal hernia or lymphadenopathy)
11. History or evidence of active tuberculosis
12. A positive QuantiFERON®-TB Gold In-Tube test
13. A household contact with active TB disease

Ages: 112 Days to 182 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 487 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, Study Director — Aeras
Locations (7):
- Kenya (3):
  - Boro Heath Center, Boro
  - KEMRI/CDC Research and Public Heath Collaboration, Kisumu
  - Siaya District Hospital, Siaya
- CISM: Centro de Investigacao em Saude de Manhica, Manhiça, Mozambique
- South Africa (3):
  - Univeristy of Cape Town, Cape Town
  - Perinatal HIV Research Unit (PHRU) Chris Hani Baragwanath Hospital, Soweto
  - SATVI: Worcester, Worcester

REFERENCES:
- [Background] Tameris M, Hokey DA, Nduba V, Sacarlal J, Laher F, Kiringa G, Gondo K, Lazarus EM, Gray GE, Nachman S, Mahomed H, Downing K, Abel B, Scriba TJ, McClain JB, Pau MG, Hendriks J, Dheenadhayalan V, Ishmukhamedov S, Luabeya AK, Geldenhuys H, Shepherd B, Blatner G, Cardenas V, Walker R, Hanekom WA, Sadoff J, Douoguih M, Barker L, Hatherill M. A double-blind, randomised, placebo-controlled, dose-finding trial of the novel tuberculosis vaccine AERAS-402, an adenovirus-vectored fusion protein, in healthy, BCG-vaccinated infants. Vaccine. 2015 Jun 9;33(25):2944-54. doi: 10.1016/j.vaccine.2015.03.070. Epub 2015 Apr 28. PMID 25936724

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Finding - Group 1: Subjects enrolled in Study Group 1 will receive two doses of placebo once on Study Day 0 and again on Study Day 28.
  Placebo: Sterile buffer
- Dose Finding - Group 2: Subjects enrolled in Study Group 2 will receive two doses of AERAS-402 (1.5 x 10^10 vp) once on Study Day 0 and again on Study Day 28.
  AERAS-402 1.5 x 10^10 vp: Live recombinant serotype 35 replication deficient adenovirus vector expressing a fusion protein of three Mycobacterium tuberculosis antigens.
- Dose Finding - Group 3: Subjects enrolled in Study Group 3 will receive two doses of AERAS-402 (3.0 x 10^10 vp) once on Study Day 0 and again on Study Day 28.
  AERAS-402 3.0 x 10^10 vp: Live recombinant serotype 35 replication deficient adenovirus vector expressing a fusion protein of three Mycobacterium tuberculosis antigens.
- Dose Finding - Group 4: Subjects enrolled in Study Group 4 will receive two doses of AERAS-402 (1.0 x 10^11 vp) once on Study Day 0 and again on Study Day 28.
  AERAS-402 1.0 x 10^11 vp: Live recombinant serotype 35 replication deficient adenovirus vector expressing a fusion protein of three Mycobacterium tuberculosis antigens.
- Expanded Safety Phase - Group 5: Subjects received 3 doses of AERAS-402 (1 X 10^11 vp) on days 0, 28 and 280.
  AERAS-402 1.0 x 10^11 vp: Live recombinant serotype 35 replication deficient adenovirus vector expressing a fusion protein of three Mycobacterium tuberculosis antigens.
- Expanded Safety Phase - Group 5 Placebo: Subjects received 3 doses of placebo on days 0, 28 and 280.
  Placebo: Sterile buffer
Period: Overall Study
Arm/Group | Dose Finding - Group 1 | Dose Finding - Group 2 | Dose Finding - Group 3 | Dose Finding - Group 4 | Expanded Safety Phase - Group 5 | Expanded Safety Phase - Group 5 Placebo
Started | 52 | 51 | 51 | 52 | 140 | 141
Completed | 40 | 44 | 43 | 47 | 125 | 128
Not Completed | 12 | 7 | 8 | 5 | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Finding - Group 1 | Dose Finding - Group 2 | Dose Finding - Group 3 | Dose Finding - Group 4 | Expanded Safety Phase - Group 5 | Expanded Safety Phase - Group 5 Placebo | Total
Number analyzed (Participants) | 52 | 51 | 51 | 52 | 140 | 141 | 487
Age, Customized [Mean (Standard Deviation); unit: Days] — ≥112 days (16 weeks) and ≤182 days (26 weeks) on Study Day 0
  Days
    Age at Study Day 0 in Days | 145.3 (18.15) | 144.5 (17.83) | 138.6 (19.45) | 149.1 (21.44) | 145.2 (19.98) | 150.2 (20.22) | 146.3 (19.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 30 | 20 | 68 | 57 | 217
  Male | 30 | 31 | 21 | 32 | 72 | 84 | 270
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 42 | 44 | 41 | 43 | 102 | 98 | 370
  Coloured | 10 | 7 | 10 | 9 | 38 | 43 | 117
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Two sites in South Africa - Worcester and Soweto. Soweto only participated in Group 5.
  participants
    Mozambique | 4 | 3 | 3 | 4 | 0 | 0 | 14
    South Africa | 12 | 12 | 12 | 12 | 70 | 70 | 188
    Kenya | 36 | 36 | 36 | 36 | 70 | 71 | 285

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Collected Per Subject
Description: Adverse Events (AEs) are recorded for 28 days post vaccination Serious Adverse Events (SAEs) are recorded for the entire study period to assess the safety profile
Time Frame: Up to 24 months post vaccination
Population: Subjects who received at least one vaccination.
Measure: Number; unit: percentage of subjects with an AE
Arm/Group | Dose Finding - Group 1 | Dose Finding - Group 2 | Dose Finding - Group 3 | Dose Finding - Group 4 | Expanded Safety Phase - Group 5 | Expanded Safety Phase - Group 5 Placebo
Number analyzed (Participants) | 52 | 51 | 51 | 52 | 140 | 141
percentage of subjects with an AE | 94.2 | 96.1 | 100.0 | 100.0 | 100.0 | 98.6

2. Secondary Outcome: Percentage of Cells Expressing Various Cytokines Will be Measured by Intracellular Cytokine Staining (ICS) in All Subjects
Description: To evaluate the immunogenicity of AERAS-402 compared to controls, flow cytometric ICS of CD4 and CD8 T cells producing any of three cytokines (IFN-γ, TNF-α, and/or IL-2) alone or in combination after stimulation with a peptide pool of mycobacterial peptides. Dimethylsulfoxide (DMSO) subtracted responses are presented.
Time Frame: 28 days post last vaccination
Population: Groups 1-4: Subjects who received both vaccinations as randomized. Group 5: Subjects who received all three study vaccinations as randomized.
Measure: Median (95% Confidence Interval); unit: percentage of Tcell response
Arm/Group | Dose Finding - Group 1 | Dose Finding - Group 2 | Dose Finding - Group 3 | Dose Finding - Group 4 | Expanded Safety Phase - Group 5 | Expanded Safety Phase - Group 5 Placebo
Number analyzed (Participants) | 41 | 39 | 42 | 46 | 50 | 61
percentage of Tcell response
  Ag85A CD4 | 0.00 [0.00 to 0.00] | 0.01 [0.00 to 0.03] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.04] | 0.02 [0.01 to 0.04] | 0.00 [0.00 to 0.01]
  Ag85A CD8 | 0.00 [0.00 to 0.00] | 0.01 [0.00 to 0.04] | 0.01 [0.00 to 0.04] | 0.02 [0.00 to 0.04] | 0.04 [0.01 to 0.06] | 0.00 [0.00 to 0.01]
  Ag85B CD4 | 0.00 [0.00 to 0.01] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03] | 0.03 [0.01 to 0.04] | 0.01 [0.01 to 0.03] | 0.00 [0.00 to 0.01]
  Ag85B CD8 | 0.00 [0.00 to 0.01] | 0.04 [0.02 to 0.08] | 0.03 [0.01 to 0.05] | 0.04 [0.02 to 0.07] | 0.05 [0.03 to 0.07] | 0.00 [0.00 to 0.00]
  TB10.4 CD4 | 0.01 [0.00 to 0.01] | 0.01 [0.00 to 0.01] | 0.01 [0.00 to 0.03] | 0.01 [0.01 to 0.02] | 0.01 [0.00 to 0.01] | 0.00 [0.00 to 0.01]
  TB10.4 CD8 | 0.00 [0.00 to 0.01] | 0.01 [0.00 to 0.01] | 0.00 [0.00 to 0.01] | 0.01 [0.00 to 0.02] | 0.01 [0.00 to 0.01] | 0.00 [0.00 to 0.00]

3. Secondary Outcome: Interferon-gamma (IFN-gamma) Enzyme-linked Immunospot (ELISpot) Response: Spot Forming Units/10^6 PBMC According to ELISpot Assay
Description: To evaluate the immunogenicity of AERAS-402 compared to controls. ELISpot assay of specific T cell responses after stimulation with a peptide pool of mycobacterial peptides. Values presented have been corrected for background readings.
Time Frame: 28 days post last vaccination
Population: Groups 1 and 4: Subjects who received both vaccinations as randomized (assays were not done for Groups 2 and 3).
  Group 5: Subjects who received all three study vaccinations as randomized.
Measure: Median (95% Confidence Interval); unit: SFU/10^6 PBMC
Arm/Group | Dose Finding - Group 1 | Dose Finding - Group 2 | Dose Finding - Group 3 | Dose Finding - Group 4 | Expanded Safety Phase - Group 5 | Expanded Safety Phase - Group 5 Placebo
Number analyzed (Participants) | 26 | 0 | 0 | 34 | 43 | 46
SFU/10^6 PBMC
  Ag85A | 5.00 [2.50 to 6.67] |  |  | 87.92 [74.17 to 156.67] | 98.33 [70.00 to 151.67] | 0.00 [0.00 to 3.33]
  Ag85B | 0.42 [0.00 to 5.00] |  |  | 127.08 [70.83 to 285.00] | 65.00 [51.67 to 133.33] | 0.83 [0.00 to 5.00]
  TB10.4 | 5.42 [0.83 to 11.67] |  |  | 26.67 [19.17 to 49.17] | 17.50 [11.67 to 28.33] | 3.33 [1.67 to 6.67]

4. Secondary Outcome: Antigen-specific Antibody Response - Mean Optical Density (Mean OD)
Description: To evaluate the immunogenicity of AERAS-402 compared to controls by ELISA Assay for Antigen-specific Antibody Response. Median responses of individual Mean OD (absorbance at 450nm) by study group is presented. Higher OD values suggests the presence of antibody to each of the Mtb antigens (Ag85A, Ag85B and TB10.4).
Time Frame: 28 day post last vaccination
Population: Groups 1 and 4: Subjects who received both vaccinations as randomized (assays were not done for Ag85A and TB10.4).
  Assays were not done for groups 2 and 3 for any antigen. Group 5: Subjects who received all three study vaccinations as randomized.
Measure: Median (95% Confidence Interval); unit: Optical Density
Arm/Group | Dose Finding - Group 1 | Dose Finding - Group 2 | Dose Finding - Group 3 | Dose Finding - Group 4 | Expanded Safety Phase - Group 5 | Expanded Safety Phase - Group 5 Placebo
Number analyzed (Participants) | 19 | 0 | 0 | 32 | 18 | 16
Optical Density
  Ag85A | NA [NA to NA] — This group was not analyzed. |  |  | NA [NA to NA] — This group was not analyzed. | 1.34 [1.08 to 2.37] | 0.20 [0.14 to 0.30]
  Ag85B | 0.26 [0.12 to 0.38] |  |  | 2.15 [1.80 to 2.53] | 2.17 [1.95 to 3.04] | 0.37 [0.28 to 0.72]
  TB10.4 | NA [NA to NA] — This group was not analyzed. |  |  | NA [NA to NA] — This group was not analyzed. | 0.94 [0.39 to 1.50] | 0.34 [0.25 to 0.46]

5. Secondary Outcome: Percentage of Subjects Converting From a Negative QuantiFERON Test (QFT) to Positive QFT After Vaccination
Description: To evaluate the proportion of on-study QuantiFERON conversions from negative to positive in infants that received AERAS-402 compared to controls. A QFT value of on >= 0.35IU/mL was considered positive for this study.
Time Frame: up to 24 months post vaccination
Population: Subjects who received at least one vaccination and had results at baseline and end of study.
Measure: Number; unit: % converting from QFT neg to pos
Arm/Group | Dose Finding - Group 1 | Dose Finding - Group 2 | Dose Finding - Group 3 | Dose Finding - Group 4 | Expanded Safety Phase - Group 5 | Expanded Safety Phase - Group 5 Placebo
Number analyzed (Participants) | 38 | 44 | 43 | 47 | 124 | 128
% converting from QFT neg to pos | 0 | 13.6 | 0 | 4.3 | 2.4 | 4.7

ADVERSE EVENTS:
Time Frame: Up to 24 months
Groups:
- Dose Finding - Group 1: Subjects received two doses of placebo (sterile buffer) on study days 0 and 28.
- Dose Finding - Group 2: Subjects received two doses of AERAS-402 (1.5 x 10^10 vp) on study days 0 and 28.
- Dose Finding - Group 3: Subjects received two doses of AERAS-402 (3.0 x 10^10 vp) on study days 0 and 28.
- Dose Finding - Group 4: Subjects received two doses of AERAS-402 (1.0 x 10^11 vp) on study days 0 and 28.
- Expanded Safety Phase - Group 5: Subjects received 3 doses of AERAS-402 (1.0 X 10^11 vp) on days 0, 28 and 280.
- Expanded Safety Phase - Group 5 Placebo: Subjects received 3 doses of placebo (sterile buffer) on days 0, 28 and 280.
  Placebo
Arm/Group | Dose Finding - Group 1 | Dose Finding - Group 2 | Dose Finding - Group 3 | Dose Finding - Group 4 | Expanded Safety Phase - Group 5 | Expanded Safety Phase - Group 5 Placebo
Serious Adverse Events (participants affected / at risk) | 20/52 | 25/51 | 23/51 | 18/52 | 40/140 | 38/141
Other Adverse Events (participants affected / at risk) | 48/52 | 47/51 | 49/51 | 52/52 | 136/140 | 139/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Finding - Group 1 (N=52) | Dose Finding - Group 2 (N=51) | Dose Finding - Group 3 (N=51) | Dose Finding - Group 4 (N=52) | Expanded Safety Phase - Group 5 (N=140) | Expanded Safety Phase - Group 5 Placebo (N=141)
Bronchiolitis (Infections and infestations) | 2 (2) | 1 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Burn infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (3) | 7 (7) | 4 (4) | 8 (8) | 11 (14)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 12 (16) | 18 (22) | 11 (13) | 8 (12) | 14 (16) | 12 (18)
Measles (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (12) | 7 (9) | 6 (6) | 6 (6) | 11 (13) | 5 (5)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salmonella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal scalded skin syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Finding - Group 1 (N=52) | Dose Finding - Group 2 (N=51) | Dose Finding - Group 3 (N=51) | Dose Finding - Group 4 (N=52) | Expanded Safety Phase - Group 5 (N=140) | Expanded Safety Phase - Group 5 Placebo (N=141)
Bronchiolitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 4 (5) | 2 (3)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 9 (14) | 12 (12)
Gastroenteritis (Infections and infestations) | 6 (6) | 4 (4) | 4 (4) | 10 (11) | 24 (25) | 20 (21)
Malaria (Infections and infestations) | 13 (14) | 18 (21) | 17 (21) | 17 (22) | 34 (50) | 35 (48)
Measles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 9 (9)
Oral candidiasis (Infections and infestations) | 4 (4) | 5 (5) | 3 (4) | 2 (2) | 5 (6) | 3 (3)
Pneumonia (Infections and infestations) | 13 (20) | 7 (7) | 8 (12) | 18 (25) | 26 (30) | 20 (21)
Rhinitis (Infections and infestations) | 3 (3) | 2 (2) | 4 (5) | 8 (8) | 6 (7) | 6 (6)
Tinea capitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 31 (47) | 32 (46) | 36 (55) | 37 (55) | 117 (248) | 114 (214)
Urinary tract infection (Infections and infestations) | 6 (7) | 3 (3) | 4 (4) | 5 (5) | 16 (16) | 19 (19)
Lymphadenopathy (Blood and lymphatic system disorders) | 6 (6) | 6 (7) | 4 (6) | 6 (6) | 47 (77) | 48 (70)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 5 (5) | 0 (0)
Conjunctivitis (Eye disorders) | 5 (5) | 8 (9) | 12 (13) | 10 (10) | 30 (36) | 20 (26)
Eye discharge (Eye disorders) | 2 (2) | 2 (3) | 4 (6) | 1 (1) | 3 (3) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 4 (5) | 4 (6) | 4 (5) | 3 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 7 (7) | 1 (1) | 4 (5) | 4 (4)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 32 (51) | 28 (52) | 31 (51) | 30 (42) | 61 (102) | 56 (96)
Diarrhoea (Gastrointestinal disorders) | 29 (49) | 30 (53) | 30 (50) | 28 (46) | 87 (151) | 71 (103)
Vomiting (Gastrointestinal disorders) | 5 (6) | 11 (11) | 6 (7) | 1 (1) | 7 (7) | 1 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 1 (1) | 2 (2) | 12 (12) | 15 (16)
Rash (Skin and subcutaneous tissue disorders) | 13 (17) | 11 (12) | 12 (13) | 9 (9) | 28 (32) | 39 (48)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 3 (3) | 3 (3) | 1 (1) | 3 (3)
Fatigue (General disorders) | 8 (10) | 8 (8) | 12 (12) | 16 (19) | 40 (59) | 16 (22)
Feeling hot (General disorders) | 4 (4) | 4 (5) | 5 (5) | 16 (20) | 37 (43) | 18 (19)
Hypothermia (General disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 3 (5) | 4 (4) | 11 (13) | 30 (42) | 5 (5)
Injection site pain (General disorders) | 6 (7) | 15 (17) | 24 (28) | 37 (54) | 104 (191) | 23 (28)
Injection site swelling (General disorders) | 6 (6) | 14 (19) | 9 (9) | 17 (22) | 46 (60) | 12 (14)
Pyrexia (General disorders) | 3 (3) | 6 (6) | 7 (7) | 13 (13) | 60 (76) | 19 (22)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 9 (10) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 3 (3) | 9 (10)
Blood bilirubin increased (Investigations) | 14 (15) | 12 (12) | 19 (20) | 12 (16) | 35 (37) | 28 (34)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 13 (15) | 9 (10)
Haemoglobin decreased (Investigations) | 12 (15) | 9 (9) | 9 (9) | 19 (19) | 36 (38) | 32 (37)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 8 (10)
Lymphocyte count increased (Investigations) | 11 (11) | 12 (12) | 16 (16) | 9 (9) | 8 (8) | 8 (8)
Neutrophil count decreased (Investigations) | 6 (6) | 7 (7) | 4 (4) | 7 (8) | 18 (20) | 21 (24)
Platelet count decreased (Investigations) | 3 (3) | 1 (1) | 2 (3) | 3 (3) | 6 (6) | 9 (9)
Platelet count increased (Investigations) | 7 (7) | 10 (10) | 10 (10) | 7 (7) | 11 (11) | 3 (3)
Protein urine (Investigations) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 4 (5) | 8 (8)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 11 (11)
White blood cell count increased (Investigations) | 4 (4) | 1 (1) | 5 (5) | 0 (0) | 3 (3) | 6 (6)
White blood cells urine (Investigations) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No